CLINICAL TRIAL: NCT03152591
Title: A Randomized, Subject- and Investigator-blinded, Placebo-controlled Pharmacodynamic Study of Oral LIK066 in Overweight and Obese Women With Polycystic Ovary Syndrome
Brief Title: Study of Pharmacodynamics of LIK066 in Overweight and Obese Women With Polycystic Ovary Syndrome
Acronym: PCOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CLIK066X2205; 2017-001373-16 (EudraCT Number)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Results first posted 2019-05-09 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; PCOS; hyperandrogenism; insulin resistance; overweight; obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Insulin Resistance; Overweight; Obesity | interventions — licogliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LIK066 (Experimental): LIK066 tablets received three times daily; before breakfast, lunch and dinner for 14 days and once on day 15 morning before meal test
  Interventions: Drug: LIK066
- Placebo (Placebo Comparator): Placebo tablets received three times daily; before breakfast, lunch and dinner for 14 days and once on day 15 morning before meal test
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIK066 — LIK066 tablets for oral administration
  Arms: LIK066
Drug: Placebo — Placebo tablets matching LIK066 tablets, for oral administration
  Arms: Placebo

SUMMARY:
The purpose of the study was to evaluate whether LIK066 can be developed for the treatment of polycystic ovary syndrome (PCOS) in overweight and obese women.

ELIGIBILITY:
Key Inclusion Criteria:

* PCOS (diagnosed as clinical or biochemical hyperandrogenism, amenorrhea or oligomenorrhea and exclusion of other causes of hyperandrogenism.
* Overweight/obese female subjects with BMI of 28 - 45 kg/m^2, inclusive, and stable weight +/- 3 kg over previous 3 months
* Subjects must use non-hormonal methods of contraception during the study.

Key Exclusion Criteria:

* Subjects with exogenous causes of hirsutism
* Menstruation in the 30 days prior to screening or treatment
* Pregnant or nursing (lactating) women
* Use of prohibited medications
* Preexisting medical condition which may significantly alter the absorption, metabolism, or excretion of the study drug, or which may jeopardize the subject in case of participation in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (2):
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 5 centers in 2 countries: Germany (3), and USA (2).
Pre-assignment Details: Participants were randomized in the ratio of 1:1 to receive either LIK066 50 mg tid or placebo for 14 days and morning dose on Day 15.
Period: Overall Study
Arm/Group | LIK066 | Placebo
Started (All randomized patients were included in the Full Analysis Set (FAS) and Safety Analysis Set (SAF).) | 15 | 14
Pharmacokinetic (PK) Analysis Set (At least one dose of study drug and one evaluable PK concentration measurement) | 14 | 0
Pharmacodynamic (PD) Analysis Set (At least one dose of study drug and one evaluable PD assessment) | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LIK066 | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.1 (4.76) | 29.1 (5.66) | 27.6 (5.34)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 15 | 14 | 29
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 15 | 14 | 29
Average fasting total testosterone [Mean (Standard Deviation); unit: nmol/L] | 1.98 (0.841) | 2.07 (0.608) | 2.02 (0.724)
Average fasting free testosterone [Mean (Standard Deviation); unit: nmol/L] | 0.037 (0.0163) | 0.032 (0.0086) | 0.034 (0.0132)
Sex hormone binding globulin (SHBG) [Mean (Standard Deviation); unit: nmol/L] | 18.3 (7.72) | 24.6 (10.51) | 21.4 (9.58)
Free androgen Index [Mean (Standard Deviation); unit: ratio] — Free Androgen Index (FAI) is a ratio used to determine abnormal androgen status in humans. The ratio is the total testosterone level divided by the sex hormone binding globulin (SHBG) level, and then multiplying by 100. FAI has no units.
  ratio | 12.4 (6.65) | 9.0 (2.77) | 10.7 (5.27)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Morning Fasting Free Testosterone Blood Concentrations From Baseline
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: nmol/L
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
nmol/L | 0.91 [0.77 to 1.07] | 1.03 [0.88 to 1.21]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.353, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ratio LIK066/Placebo = 0.88, 90% CI 2-sided [0.70 to 1.11]; Log transformed ratio of Day 15 to baseline in average fasting free testosterone was analyzed using an analysis of covariance model which included treatment as a categorical factor, baseline body weight and log transformed baseline average fasting free testosterone as a covariate

2. Secondary Outcome: Change From Baseline in Luteinizing Hormone (LH) at Day 15
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: U/L
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
U/L | 1.37 [1.11 to 1.69] | 1.10 [0.89 to 1.36]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.218, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ratio LIK066/Placebo = 1.25, 90% CI 2-sided [0.92 to 1.68]; Log transformed ratio of Day 15 to baseline was analyzed using an analysis of covariance model which will include treatment as a categorical factor and log transformed baseline as a covariate

3. Secondary Outcome: Change From Baseline in Follicle Stimulating Hormone (FSH) at Day 15
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: U/L
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
U/L | 1.13 [0.89 to 1.43] | 0.89 [0.70 to 1.13]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.249, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ratio LIK066/Placebo = 1.27, 90% CI 2-sided [0.90 to 1.78]; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Sex Hormone Binding Globulin (SHBG) at Day 15
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: nmol/L
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
nmol/L | 1.06 [0.95 to 1.20] | 0.93 [0.83 to 1.03]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.173, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ratio LIK066/Placebo = 1.15, 90% CI 2-sided [0.97 to 1.36] — Values < LLOQ and values > ULOQ are imputed as LLOQ/2 and ULOQ respectively; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in Androstenedione at Day 15
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: nmol/L
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
nmol/L | 0.85 [0.74 to 0.97] | 1.03 [0.91 to 1.17]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.089, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ratio LIK066/Placebo = 0.82, 90% CI 2-sided [0.68 to 0.99] — Values < LLOQ and values > ULOQ are imputed as LLOQ/2 and ULOQ respectively; [other analysis details as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline in Dehydroepiandrostenedione (DHEA) at Day 15
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: nmol/L
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
nmol/L | 0.75 [0.58 to 0.98] | 1.09 [0.85 to 1.39]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.109, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ration LIK066/Placebo = 0.69, 90% CI 2-sided [0.48 to 1.01] — Values < LLOQ and values > ULOQ are imputed as LLOQ/2 and ULOQ respectively; [other analysis details as in outcome 2, analysis 1]

7. Secondary Outcome: Change From Baseline in Dehydroepiandrostenedione Sulfate (DHEAS) at Day 15
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: umol/L
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
umol/L | 0.84 [0.75 to 0.94] | 1.10 [0.99 to 1.23]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.008, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ration LIK066/Placebo = 0.76, 90% CI 2-sided [0.65 to 0.89] — Values < LLOQ and values > ULOQ are imputed as LLOQ/2 and ULOQ respectively; [other analysis details as in outcome 2, analysis 1]

8. Secondary Outcome: Change From Baseline in Total Testosterone, at Day 15
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: nmol/L
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
nmol/L | 0.95 [0.84 to 1.06] | 1.04 [0.92 to 1.17]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.340, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ratio LIK066/Placebo = 0.91, 90% CI 2-sided [0.77 to 1.07]; [other analysis details as in outcome 2, analysis 1]

9. Secondary Outcome: Change From Baseline in Free Androgen Index (FAI), at Day 15
Description: Free Androgen Index (FAI) is a ratio used to determine abnormal androgen status in humans. The ratio is the total testosterone level divided by the sex hormone binding globulin (SHBG) level, and then multiplying by 100. FAI has no units.
Time Frame: Baseline, Day 15
Population: Pharmacodynamic (PD) analysis set
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | LIK066 | Placebo
Number analyzed (Participants) | 15 | 14
Ratio | 0.85 [0.69 to 1.05] | 1.07 [0.88 to 1.31]
Statistical Analysis 1: Comparison: LIK066 vs Placebo; Test type: Other; p = 0.204, t-test, 2 sided; Two-sided test at the 0.1 significance level; Ratio LIK066/Placebo = 0.79, 90% CI 2-sided [0.58 to 1.08] — Values < LLOQ and values > ULOQ are imputed as LLOQ/2 and ULOQ respectively; [other analysis details as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the maximum duration of participants' treatment exposure plus any follow up period, approximately 2 months.
Arm/Group | LIK066 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 15/15 | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LIK066 (N=15) | Placebo (N=14)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 15 | 3
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 6 | 0
GASTROINTESTINAL TRACT IRRITATION (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 5 | 2
VOMITING (Gastrointestinal disorders) | 0 | 1
THIRST (General disorders) | 4 | 1
NASOPHARYNGITIS (Infections and infestations) | 2 | 1
RHINITIS (Infections and infestations) | 1 | 0
VAGINAL INFECTION (Infections and infestations) | 1 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 | 0
MENSTRUATION NORMAL (Investigations) | 4 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 4 | 1
MIGRAINE (Nervous system disorders) | 0 | 1
INSOMNIA (Psychiatric disorders) | 1 | 0
MOOD ALTERED (Psychiatric disorders) | 1 | 0
POLYURIA (Renal and urinary disorders) | 0 | 1
HYPOMENORRHOEA (Reproductive system and breast disorders) | 2 | 1
MENSTRUAL DISORDER (Reproductive system and breast disorders) | 0 | 1
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT03152591/SAP_000.pdf
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03152591/Prot_001.pdf